CLINICAL TRIAL: NCT00168766
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Parallel Group Trial Investigating Methylprednisolone in Combination With Interferon-beta-1a for the Treatment of Patients With Relapsing-remitting Multiple Sclerosis
Brief Title: Avonex (Interferon-beta-1a) and Avonex Plus Methylprednisolone for the Treatment of Relapsing-remitting MS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Nordic Medical Director, Biogen Idec International
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOR-03-01; Mecombin; NCT00492180 (obsolete NCT alias)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-04

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Combination therapy for multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): interferon-beta-1a in combination with methylprednisolone
  Interventions: Drug: Interferon-beta-1a (Avonex) plus methylprednisolone
- 2 (Placebo Comparator): interferon-beta-1a in combination with placebo
  Interventions: Drug: Interferon-beta-1a (Avonex) plus methylprednisolone

INTERVENTIONS:
Drug: Interferon-beta-1a (Avonex) plus methylprednisolone — oral administration given on 3 consecutive days, monthly as described in protocol.
  Other Names: Avonex

SUMMARY:
The primary objective of this study is to determine whether combination treatment (adding methylprednisolone to Avonex) reduces progression of disability over 4 years compared to Avonex alone. The study will also investigate whether combination therapy has any impact on the incidence of relapse and brain atrophy as measured by MRI.

DETAILED DESCRIPTION:
Approximately 340 therapy-naïve MS patients with relapsing-remitting form of the disease will be randomized to receive Avonex alone or Avonex plus methylprednisolone (MP). Patients will receive MP as 500 mg po for 3 days every month or matching placebo. The patients are followed on a 3-monthly basis for 4 years with disability as the primary parameter of efficacy over that time.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Relapsing remitting MS according to Poser criteria or McDonell criteria and naïve to therapy
* Disability EDSS score of 4.0 or less at baseline
* Clinical activity as defined by at least one relapse in the last year

Exclusion Criteria:

* Relapse in the month prior to enrolment
* Treatment with immunosuppressive drugs for MS
* History of major depression
* Former severe reactions to corticosteroids
* Pregnant women
* Diabetes mellitus, and drug or alcohol dependency
* Known or suspected allergy to trial products

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2003-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To estimate the effect interferon-beta-1a in combination with methylprednisolone vs interferon-beta-1a in combination with placebo on the time to onset of disability progression sustained over at least 6 months based on change from randomization in EDSS | 4 years

CONTACTS AND LOCATIONS:
Locations (9):
- CUB Hôpital Erasme, Brussels, Belgium
- Denmark (2):
  - Coordinating Research Site, Copenhagen
  - Rigshospitalet, Skleroseklinikken
- Tampereen yliopistollinen sairaala - Neurologian klinikka, Tampere, Finland
- Stichting MS Centrum, Nijemegen, Netherlands
- Ullevål Universitetssykehus, Oslo, Norway
- Neurologkliniken, Stockholm, Sweden
- Kantonspital, Sankt Gallen, Switzerland
- Queens Medical Centre - Division of Neurology, Nottingham, United Kingdom

REFERENCES:
- [Derived] Ravnborg M, Sorensen PS, Andersson M, Celius EG, Jongen PJ, Elovaara I, Bartholome E, Constantinescu CS, Beer K, Garde E, Sperling B. Methylprednisolone in combination with interferon beta-1a for relapsing-remitting multiple sclerosis (MECOMBIN study): a multicentre, double-blind, randomised, placebo-controlled, parallel-group trial. Lancet Neurol. 2010 Jul;9(7):672-80. doi: 10.1016/S1474-4422(10)70132-0. Epub 2010 Jun 9. PMID 20542736